CLINICAL TRIAL: NCT05531838
Title: A Community Controlled Study of MMC Mode Combined With CGM Therapeutic Monitoring Technology in the Management of Patients With Prediabetes
Brief Title: Prediabetes Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Liping Gu, associate chief physician, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CTCCR-2021C20
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: PreDiabetes; Metabolic Management Center; Continuous Glucose Monitoring
Keywords: prediabetes; continuous glucose monitoring; metabolic management center
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fu Lishan instant sense hospital dynamic glucose monitoring system (Other): Using CGM Technology (dynamic glucose monitoring system for Fu Lishan instant sense hospital), on the basis of the original eating habits of patients, according to the guidelines and the training of MMC center, patients are guided to adjust the diet model according to the glucose map monitored by the dynamic glucose monitoring system and the log recorded, so as to implement therapeutic monitoring, control the blood glucose level within the target range as far as possible, and record the amount of various foods accordingly, After that, the eating method and amount remained basically unchanged.
  Interventions: Device: Fu Lishan instant sense hospital dynamic glucose monitoring system

INTERVENTIONS:
Device: Fu Lishan instant sense hospital dynamic glucose monitoring system — Using CGM Technology (dynamic glucose monitoring system used in Fu Lishan instant sense hospital), on the basis of patients' original eating habits, according to the guidelines and the training of MMC center, patients are guided to adjust their eating patterns according to the glucose map monitored by the dynamic glucose monitoring system.

SUMMARY:
Systematically screen the high-risk population of diabetes in Xinqiao district to understand the characteristics of early glucose metabolism changes and pancreatic islet function changes in patients with pre diabetes. Relying on MMC platform and combined with CGM therapeutic monitoring technology to standardize the management of patients with prediabetes, it is expected that the annual conversion rate of diabetes in patients with prediabetes will be 8% (according to the literature, if the pre diabetes population is not intervened, the annual conversion rate of diabetes will be about 14%), which will move forward the management of diabetes and create a new mode of pre diabetes management.

DETAILED DESCRIPTION:
Part I: Establish the first standardized study cohort of prediabetes patients in Songjiang

On the basis of previous studies, we will continue to carry out early screening of diabetes high-risk groups. It is planned to complete 500 high-risk screening cases in Xinqiao area, and all screened patients will have their medical history and relevant laboratory examinations, and will be followed up regularly. The standard OGTT method was used for screening. The screening contents included: fasting blood glucose and insulin, blood glucose and insulin levels 2 hours after 75g glucose load, and glycosylated hemoglobin levels. In addition to glucose metabolism, other metabolic related diseases such as hematuria routine, liver and kidney function, uric acid, blood lipids, thyroid function, and urine protein / creatinine were also screened. The establishment of the high-quality high-risk screening project in Xinqiao community will establish the first standardized research cohort of diabetes high-risk and pre diabetes patients in Songjiang area, which has very important strategic significance.

Part II: Standardized management and follow-up based on MMC mode combined with CGM therapeutic monitoring technology

For patients with pre diabetes diagnosed by screening, we will rely on MMC mode and CGM technology for standardized management and follow-up. The management mode is mainly embodied in the following forms: ① using CGM Technology (dynamic glucose monitoring system for auxiliary Lishan instant sense hospital), on the basis of the original eating habits of patients, according to the guidelines and the training of MMC center, patients are guided to adjust their eating mode according to the glucose map monitored by the dynamic glucose monitoring system and the log recorded, so as to implement therapeutic monitoring, so as to control the blood glucose level within the target range as far as possible, And record the amount of various foods accordingly, and then maintain the eating mode and amount basically unchanged. ② Offline management. Patient education at least twice a year and hospital follow-up once a year; ③ Issue health instruction manuals, blood glucose monitoring diaries, etc; ④ A full-time wechat management group is established, and full-time intelligent assistants push diet, sports and other guidance every day. Taking the cases of diabetes patients screened in the previous study of the research group as the control, the annual conversion rate of diabetes was observed one year later.

ELIGIBILITY:
Inclusion Criteria:

* IConforms to the pre diabetes in the diagnostic criteria of type 2 diabetes in the Chinese guidelines for the prevention and treatment of type 2 diabetes (version 2020) (only use plasma glucose at 0 minutes in OGTT and 120 minutes after taking glucose);

  * Initial screening and diagnosis; ③ without other serious basic diseases; ④ Have complete cognition, reading and writing ability, have a smart phone, can use simple functions, and know how to use wechat; ⑤ Those who voluntarily participate in this study are willing to sign the informed consent form.

Exclusion Criteria:

* Those who have been diagnosed with diabetes;

  * Patients with severe heart, lung, liver and kidney dysfunction;

    * Those with mental disorder, language disorder or senile dementia; ④ Those who can't take care of themselves, are bedridden or have mobility problems; ⑤ Lactating or pregnant women; ⑥ Patients with recent history of surgery, trauma, cardio cerebral and other acute large vessel complications and infectious diseases.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-10-17 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of diabetes | one year
  Incidence rate of patients with pre diabetes turning into diabetes after one year of standardized management

SECONDARY OUTCOMES:
HbA1c increased by 0.5% | one year
  HbA1c increased by 0.5%